CLINICAL TRIAL: NCT01670903
Title: the Effect of Angiotensin II Type 1 Receptor Antagonists on the Size and Expansion Rate of Abdominal Aortas in Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Daniel Silverberg, Senior consultant - Vascular surgery, Sheba Medical Center
Other Study IDs: SHEBA-12-8336-DS-CTIL
Record Dates: First submitted 2012-08-19; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Aneurysm; Hypertension
MeSH Terms: conditions — Aneurysm; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ARBs: Hypertensive patients treated with ARBs
- ACE inhibitors: Hypertensive patients treated with ACE inhibitors
- non ARB/ACE: Hypertensive patients treated with non ARBs or ACE inhibitors meds

SUMMARY:
Abdominal aortic aneurysm (AAA) is a common disease that develops from degeneration of the aortic wall. The natural history of AAA is gradual expansion and if left untreated may result in rupture and death. The mechanism of the development of this disease is unknown however it appears to be multifactorial and possibly related to degradation processes within the arterial wall. There is growing evidence that Angiotensin receptor blockers ( ARBS) may have an inhibitory effect on remodelling processes within the arterial wall, thus inhibiting degeneration of the vessel wall.

Study hypothesis: ARBS are associated with smaller diameters of aortas among hypertensive patients, and are associated with a lower rate of aortic expansion compared to other antihypertensive drugs.

ELIGIBILITY:
Inclusion Criteria:

* medically treated hypertensive patients, ages 50-80

Exclusion Criteria:

* pregnant women
* patients previously treated for aortic disease
* unable to sign informed consent, minors

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medically treated hypertensive patients, ages 50-80
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-05

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Silverberg, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel